CLINICAL TRIAL: NCT01841840
Title: The Acute Effects of Passive Vibration on Cardiovascular Function in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012.7712
Record Dates: First submitted 2013-04-23; First posted 2013-04-29 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Stroke; Hemiparesis; Pre-Hypertension; Hypertension
Keywords: Stroke; Hemiparetic; Passive Vibration; Arterial Stiffness; Pulse Wave Velocity; Wave Reflection; Body Composition; Autonomic Function
MeSH Terms: conditions — Stroke; Paresis; Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): This arm involves not implementing any form of intervention (passive vibration)on the subject during this visit.
- Low-Frequency Pasive Vibration (Experimental): This arm involves exposing the subject to a 10 minute session of passive vibration set to a frequency of 25Hz and a high amplitude.
  Interventions: Other: Low-Frequency Passive Vibration
- High-Frequency Passive Vibration (Experimental): This arm involves exposing the subject to a 10 minute session of passive vibration set to a frequency of 40Hz and a low amplitude.
  Interventions: Other: High-Frequency Pasive Vibration

INTERVENTIONS:
Other: Low-Frequency Passive Vibration — 10 minute session of passive vibration set to a frequency of 25Hz and a high amplitude exposed to the legs
  Other Names: Power Plate Pro5 AIRdaptive
  Arms: Low-Frequency Pasive Vibration
Other: High-Frequency Pasive Vibration — 10 minute session of passive vibration set to a frequency of 40Hz and a low amplitude exposed to the legs
  Other Names: Power Plate Pro5 AIRdaptive
  Arms: High-Frequency Passive Vibration

SUMMARY:
Stroke is the third leading cause of death in the United States. Of those who are affected by stroke, a third becomes permanently disabled. Risk factors for stroke include, but are not limited to, advancing age, physical inactivity, arterial stiffness, and most commonly, high blood pressure. Stroke is a major form of a much boarder problem, cardiovascular disease (CVD). CVD is considered the primary cause of death in the US. Interestingly, increased arterial stiffness of elastic arteries (carotid and aorta) has been shown to be strongly correlated to CVD and stroke. Increased arterial stiffness is considered an independent risk for the development of CVD and stroke. Hence, arterial stiffness has been suggested as a potential therapeutic target for CVD and more specifically stroke.

Recently, whole-body vibration (WBV) exercise has been proposed as a new and effective method to improve muscle mass and muscle strength in younger and older individuals. It is known that systemic arterial stiffness decreased 40 min after a single WBV session in healthy men. In our laboratory, we have shown that leg arterial stiffness decreases after a session of WBV. Taken together, this data seems to suggest WBV may be used as a viable way to decrease arterial stiffness. Special populations, such as post-stroke patients, may be unwilling or unable to perform WBV exercise so an inactive form of exercise (vibration) therapy is needed.

Passive vibration (PV), allows patients to lie in an inactive, supine position, with their legs placed onto the vibration plate. This exposes the lower limbs to continuous vibration without performing voluntary muscle contraction. PV has been shown to increase skin blood flow on the vibrated extremity through vasodilation in healthy individuals and type 2 diabetics. Previous work in our laboratory has demonstrated that a 10-min session of PV on the legs decreases augmentation index (AIx) , a marker of pressure wave reflection, as well as leg and systemic PWV through decreases in local peripheral resistance in young men. However, the effects of PV on arterial function in post-stroke patients are unknown.

It is hypothesized that post-stroke patients will demonstrate a decrease in leg PWV and central AIx. However, greater responses are expected with the lower vibration frequency.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of one acute bout of low and high frequency passive vibration on blood pressure, heart rate, arterial stiffness, wave reflection, and autonomic function in post-stroke patients.

The specific aim of this study is:

-To evaluate the effects of an acute bout of both high (40Hz/low amplitude) and low frequency (25Hz/high amplitude) passive vibration on arterial function and aortic hemodynamics by assessing blood pressures (systolic, diastolic, mean, pulse pressure), arterial stiffness (aortic, systemic, leg), aortic wave reflection (augmentation index), and autonomic function (heart rate variability).

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* Resting Blood Pressure between 120/80 and 159/99
* Non-Smoker
* Sedentary or low activity (<120 min per week)
* 25-39.9 kg/m2 BMI
* Diagnosed with stroke for at least 4 months

Exclusion Criteria:

* Younger than 40 and older than 80 years of age
* Resting Blood Pressure below 120/80 or above 159/99
* Smoker
* Physically active
* BMI below 25 kg/m2 or above 39.9 kg/m2
* Diagnosed with stroke for less than 4 months
* Diagnosed with any other cardiovascular diseases besides stroke and stage-1 hypertension

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressures | 30 minutes
  Non-invasive measures of brachial blood pressure
Arterial Stiffness | 30 minutes
  Using pulse wave velocity of the aorta, systemic, and legs
Pressure Wave Reflection | 30 minutes
  Using the augmentation index from radial tonometry

SECONDARY OUTCOMES:
Body Composition | 30 minutes
  By measuring fat mass and lean soft tissue mass from dual-energy x-ray absorptiometry and waist circumference
Autonomic Function | 30 minutes
  Heart rate variability will be assessed from electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, M.D., Ph.D, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States